CLINICAL TRIAL: NCT02736201
Title: Mechanosensitivity, Morphological, Functional and Contractility Changes by the Capacitive Diathermy in Subjects With Lumbopelvic Pain: a Pilot Study, Single Blind, Randomized Controlled Clinical Trial
Brief Title: Capacitive Diathermy in the Lumbopelvic Pain
Acronym: T-Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European University of Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIPI/054/15
Record Dates: First submitted 2016-03-24; First posted 2016-04-13 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMT+ T-CaRe®on; n = 10 (Experimental): The instrumental manual therapy with the switched on capacitive diathermy electrode
  Interventions: Device: Capacitive diathermy (T-CaRe®); Other: Instrumental manual therapy
- IMT+ T-CaRe® off; n = 10 (Sham Comparator): The instrumental manual therapy with the switched off capacitive diathermy electrode
  Interventions: Device: Capacitive diathermy (T-CaRe®); Other: Instrumental manual therapy

INTERVENTIONS:
Device: Capacitive diathermy (T-CaRe®) — The instrumental manual therapy with the switched on capacitive diathermy electrode (IMT+ T-CaRe® on; n = 10) and the instrumental manual therapy with the switched off capacitive diathermy electrode (IMT+ T-CaRe® off; n = 10) will be bilaterally treated for 4 weeks (1 treatment per week during 10 minutes) in the lumbopelvic region.
Other: Instrumental manual therapy — Bilateral longitudinal massage in the lumbar region (110 mm; 5 minutes in each side)

SUMMARY:
Objective: To determine the effectiveness of the capacitive diathermy in the mechanosensitivity, morphological, functional and contractility changes in patients with lumbopelvic pain.

Design: A pilot study, single blind, randomized controlled clinical trial, approved previously by The Princess University Hospital Ethics Committee (Feb 11, 2016) and the European University clinical intervention review board (CIPI/054/15).

Setting: Faculty of Health Sciences, Exercise and Sport. European University of Madrid.

Patients and intervention: A sample of 20 patients with bilateral lumbopelvic pain, between 18 and 60 years old, will be recruited and randomized into 2 intervention groups. The instrumental manual therapy with the switched on capacitive diathermy electrode (IMT+ T-CaRe®on; n = 10) and the instrumental manual therapy with the switched off capacitive diathermy electrode (IMT+ T-CaRe®off; n = 10) will be bilaterally treated for 4 weeks (1 treatment per week during 10 minutes) in the lumbopelvic region.

Outcome measurements: Control variables such as the age, sex, height, weight, body mass index, Borg scale physical activity and distress respiratory test will be measured at the beginning of the treatment. Dependent variables such as the pain intensity, the pressure pain threshold, the contractility, the stiffness, the adverse effects, the Oswestry and Schöber test, as well as the ultrasound imaging cross sectional area and thickness of the skin, subcutaneous tissue, connective tissue, L4 multifidus and the abdominal Wall (rectus anterior, externus oblique, internal oblique and transversus abdominis) will be assessed before and after each intervention by a blinded examiner.

Analysis data: The statistical analysis will be performed with a 95% confidence interval and the Statistic Package Social Sciences (SPSS) 22.0.

ELIGIBILITY:
Inclusion Criteria:

* bilateral lumbopelvic pain for 6 weeks

Exclusion Criteria:

* neuromuscular conditions
* negative straight leg raise test
* respiratory or congenital conditions
* surgeries
* neurologic signs
* lower extremities conditions
* skin alterations
* cognitive disorders
* body mass index higher than 31 kg/cm2
* skin alterations
* pregnancy
* intensive physical activity
* Nijmegen test higher than 24

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity from 0 to 10 | 4 weeks
  Visual analogue scale

SECONDARY OUTCOMES:
Pressure pain threshold in kg/cm^2 | 4 weeks
  Analogue pressure algometer (Mechanical algometer)
Contractility time in seconds | 4 weeks
  Electrical stimulator
Stiffness by the mean strain ratio (proportion) by Sonoelastography | 4 weeks
  The mean strain ratio by Sonoelastography
Adverse effects (yes or no) | 4 weeks
Oswestry test from 0 to 100 | 4 weeks
Schöber test in centimeters | 4 weeks
Cross sectional area (cm^2) in centimeters | 4 weeks
  Ultrasound imaging (cm^2) in the L4 multifidus of the low back region and the rectus anterior of the abdominal wall. Diagnostic ultrasound system.
Thickness in centimeters | 4 weeks
  Ultrasound imaging (cm) in the skin, subcutaneous tissue, connective tissue, L4 multifidus and the abdominal Wall (rectus anterior, external oblique, internus oblique and transversus abdominis). Diagnostic ultrasound system

OTHER OUTCOMES:
Age in years. | 1 day
Sex (men / women) | 1 day
height in meters | 1 day
weight in kilograms | 1 day
body mass index in kg/m^2 | 1 day
Borg physical scale from 0 to 10 | 1 day
Nijmegen distress respiratory test from 0 to 64 | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: César Calvo Lobo, PhD, MSc, PT, Principal Investigator — European University of Madrid; David Rodríguez Sanz, PhD, MSc, PT, Principal Investigator — European University of Madrid
Locations (1):
- European University of Madrid, Villaviciosa de Odón, Madrid, Spain